CLINICAL TRIAL: NCT00284219
Title: High-Frequency Repetitive Transcranial Magnetic Stimulation Assists In Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Revital Amiaz, MD - Senior psychiatrist, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-04-3401-RA-CTIL
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Heavy Smoking
Keywords: rTMS, smoking, dopamine, acotinine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Real high frequency rTMS (Active Comparator): The patients will undergo a series of treatments of high frequency rTMS
  Interventions: Device: Transcranial Magnetic Stimulation 10Hz
- Sham high frequency rTMS (Sham Comparator): The patients will receive a series of sham treatments.
  Interventions: Device: Magnetic stimulation using a special sham coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation 10Hz — 3. rTMS subjects will receive 20 trains of rTMS at a rate of 10 Hz for 6 seconds (1200 pulses/session). Pulses will be administered over the left dorsolateral prefrontal cortex, defined as 5 cm anterior and in a parasagital plane to the point of maximum stimulation of the abductor pollicis muscle. Pulse intensity will be set at 100% motor threshold.
  Arms: Real high frequency rTMS
Device: Magnetic stimulation using a special sham coil — Sham stimulation will be given at the same location as the active, with special sham coil.
  Arms: Sham high frequency rTMS

SUMMARY:
Cigarette smoking is a major public health problem causing significant morbidity and mortality. Yet, smoking cessation therapies are often ineffective at helping smokers break their addiction.

The mesolimbic dopaminergic reward system plays a crucial role in mediating the reinforcing effects of nicotine. Recently, acute high frequency repetitive transcranial magnetic stimulation (rTMS) of frontal brain regions has been shown to efficiently modulate the mesolimbic dopamine systems in both animals and humans. For this reason, we investigated whether 10 high-frequency (10Hz) rTMS treatments over the left dorsolateral prefrontal cortex can help people to withdraw smoking in comparison to placebo rTMS.

Smokers seeking to quit are recruited through newspaper advertisements. Participants were randomized to 10 days of either real or placebo high frequency rTMS.

ELIGIBILITY:
Inclusion Criteria:Smoking over 20 Cig a day -

Exclusion Criteria:epilepsy, psychiatry history

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
number of cigarettes smoked

CONTACTS AND LOCATIONS:
Overall Officials: Revital A Amiaz, MD, Principal Investigator — Sheba Medical Center; Abraham Zangen, Phd, Study Director — Weizmann Institute of Science
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel